CLINICAL TRIAL: NCT05086510
Title: Ablation Targets of Scar-related Ventricular Tachycardia Identified by Dynamic Functional Substrate Mapping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohammad Gamal, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASUMD83/2021
Record Dates: First submitted 2021-09-28; First posted 2021-10-21 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-07

CONDITIONS: Tachycardia, Ventricular
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sinus Rhythm (Active Comparator): This group will undergo mapping during sinus rhythm to identify and ablate late potentials that may be incriminated in the tachycardia circuit.
  Interventions: Procedure: Radiofrequency ablation
- Right ventricular extrastimulus pacing group (Active Comparator): This group will undergo mapping during right ventricular single extrastimulus pacing to identify and thus ablate potentials that might have been masked during sinus rhythm.
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — Both groups will undergo radiofrequency ablation of potentials likely responsible for the tachycardia. Those potentials are identified by the formentioned 2 distinct methods.

SUMMARY:
This study aims at comparing the recurrence rates of ventricular tachycardia ablated after being mapped by 2 different techniques.

DETAILED DESCRIPTION:
The study participants are patients presented with recurrent ventricular tachycardia.

They will be divided into 2 groups in terms of mapping. The first group will use mapping during sinus rhythm to identify late potentials that may be incriminated in the tachycardia circuit.

The other group will undergo mapping during right ventricular extrastimulus pacing to unmask hidden potentials. The identified potentials will be ablated in both groups.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with structural heart disease; previous myocardial infarction, left ventricular dilatation/systolic dysfunction, or normal left ventricular diameters/ systolic function with evidence of ventricular scar on contrast enhanced-cardiac magnetic resonance or electroanatomic map.

  * Sustained monomorphic ventricular tachycardia documented by 12-lead ECG or implantable cardioverter defibrillator (electrograms resistant to antiarrhythmic drug treatment or requiring implantable cardioverter defibrillator therapies.

Exclusion Criteria:

* • Patients with ventricular arrhythmias attributed to reversible causes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad G Elewa, Principal Investigator — AinShams university
Locations (1):
- AinShams university hospitals, Cairo, Egypt

REFERENCES:
- [Derived] Elewa MG, Altoukhy S, Badran HA, El Damanhoury H, Zarif JK. Ablation targets of scar-related ventricular tachycardia identified by dynamic functional substrate mapping. Egypt Heart J. 2023 Oct 13;75(1):87. doi: 10.1186/s43044-023-00414-w. PMID 37831212

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-DEEP Group: This group will undergo mapping during sinus rhythm to identify and ablate late potentials that may be incriminated in the tachycardia circuit.
  Radiofrequency ablation: Both groups will undergo radiofrequency ablation of potentials likely responsible for the tachycardia. Those potentials are identified by the formentioned 2 distinct methods.
- DEEP Group: This group will undergo mapping during right ventricular single extrastimulus pacing to identify and thus ablate potentials that might have been masked during sinus rhythm.
  Radiofrequency ablation: Both groups will undergo radiofrequency ablation of potentials likely responsible for the tachycardia. Those potentials are identified by the formentioned 2 distinct methods.
Period: Overall Study
Arm/Group | Non-DEEP Group | DEEP Group
Started | 20 | 20
Completed | 20 | 16
Not Completed | 0 | 4
Not completed — Lost to Follow-up | 0 | 2
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-DEEP Group | DEEP Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.75 (11.85) | 55.65 (15.87) | 54.7 (13.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 19 | 17 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of ablation points [Median (Inter-Quartile Range); unit: ablation points] | 81 [55.5 to 129.5] | 30 [22 to 44] | 47 [22 to 129.5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrence of Ventricular Tachycardia
Description: Recurrence of ventricular tachycardia implies receiving at least one appropriate implantable cardioverter defibrillator therapy or hospital admission due to symptomatic ventricular tachycardia.
Time Frame: 12 months
Population: Among the patients who completed the study, the number of patients who experienced recurrence of ventricular tachycardia after a median follow up duration of 12 months is reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-DEEP Group | DEEP Group
Number analyzed (Participants) | 20 | 20
Participants | 13 | 13

2. Secondary Outcome: Number of Participants Who Experience Cardiac Death
Description: This is defined as unexpected death where a cardiac cause is the most probable etiology
Time Frame: 12 months
Population: The number of patients who experience cardiovascular mortality after a median follow up duration of 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Non-DEEP Group | DEEP Group
Number analyzed (Participants) | 20 | 20
Participants | 5 | 4

3. Secondary Outcome: Number of Participants Who Die From Any Cause (All-cause Mortality)
Description: This includes death from any cause
Time Frame: 12 months
Population: The number of participants who die from any cause
Measure: Count of Participants; unit: Participants
Arm/Group | Non-DEEP Group | DEEP Group
Number analyzed (Participants) | 20 | 20
Participants | 5 | 4

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Non-DEEP Group | DEEP Group
All-Cause Mortality (participants affected / at risk) | 5/20 | 4/20
Serious Adverse Events (participants affected / at risk) | 3/20 | 3/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-DEEP Group (N=20) | DEEP Group (N=20)
Cardiac tamponade (Cardiac disorders) | 0 | 3
Ventricular fibrillation (Cardiac disorders) | 1 | 0
heart block (Cardiac disorders) | 1 | 0
pulmonary edema (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT05086510/Prot_SAP_000.pdf